CLINICAL TRIAL: NCT06909773
Title: The Prevalence, Disease Burden and Prognosis of COPD in Patients With Cardiovascular Diseases -A Multi-center, Prospective, Interventional Study (PRECEDE)
Brief Title: The Prevalence, Disease Burden and Prognosis of COPD in Patients With Cardiovascular Diseases
Acronym: PRECEDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: D2287L00041
Record Dates: First submitted 2025-03-12; First posted 2025-04-04 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Guideline education and implementation (Other)
  Interventions: Behavioral: Guideline education and implementation intervention

INTERVENTIONS:
Behavioral: Guideline education and implementation intervention — The intervention is implemented at the investigator level and the patient level, consisted of 3 parts：
  1. Disease education
     * Investigator level:All investigators will receive COPD and CVD disease education according to Chinese Guideline pproximately 4 weeks before the first subject is enrolled.
     * Patient level:After the subjects are enrolled, the cardiologists and pulmonologist will provide disease education on their respective disease areas,education will be provided every 4 weeks until the end of the study.
  2. Treatment:Cardiologists and pulmonologists will work together to provide treatment management for subjects with CVD and COPD.
  3. Follow-up management:the subjects will be followed up every 4 weeks.

SUMMARY:
This is a multi-center, prospective, and interventional study conducted in 3 types of cardiovascular diseases (CVD) subjects , including 3 cohorts which are patients with newly or previously diagnosed coronary heart disease ( CHD), atrial fibrillation ( AF) and chronic heart failure (CHF).

DETAILED DESCRIPTION:
The mainly purpose of this study is describe the prevalence of COPD of the subjects with 3 types of CVD who are aged 40 years or older, and also observe the effect of cardiopulmonary co management on the short term prognosis of subjects with CVD and COPD.

This study will enroll approximately 3,000 subjects, with approximately 1,000 subjects in each cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Give signed written informed consent to participate.
2. At least 40 years of age at baseline visit.
3. Previous or newly diagnosed by at least one of the 3 types of CVD which are,

   * Coronary heart disease ( CHD )
   * Atrial fibrillation (AF )
   * Chronic heart failure ( CHF )
4. Subjects have no absolute contraindications to spirometry testing.
5. Subjects have the cognitive ability to conduct questionnaires after e valuated by investigators.

Exclusion Criteria:

1. Significant diseases or conditions, which, in the opinion of the investigator, may put the subject at risk because of participation in the study or may influence either the results of the study or the subject's ability to participate in the study.
2. Women who are pregnant or lactating or are planning to become pregnant, or women of childbearing potential who are not using an acceptable method of contraception.
3. Subjects who are not able to provide written informed consent.
4. Treatment with investigational study drug or device in another clinical study within the last 30 days or five half lives prior to baseline visit , whichever is longer.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2026-10-28 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The number and percentage of COPD in subjects with CVD,CHD,AF,CHF. | Baseline
  To describe the prevalence of COPD in subjects with CVD.

SECONDARY OUTCOMES:
The hospitalization/readmission rate in subjects with COPD. | Baseline-week12
  To describe the hospitalization/readmission rate in subjects with COPD during the implementation of cardiopulmonary co-management.
The hospitalization/readmission rate in CHD, AF and CHF subjects with COPD. | Baseline-week12
  To describe the hospitalization/readmission rate in subjects with CVD during the implementation of cardiopulmonary co-management.
Change from baseline in SAQ score in subjects with CHD and COPD. | Baseline,week4,week8,week12
  To describe the effects of cardiopulmonary co-management on quality of life, symptoms and activity tolerance in subjects with COPD.
Change from baseline in AFEQT score in subjects with AF and COPD. | Baseline,week4,week8,week12
  To describe the effects of cardiopulmonary co-management on quality of life, symptoms and activity tolerance in subjects with COPD.
Change from baseline in KCCQ score in subjects with CHF and COPD. | Baseline,week4,week8,week12
  To describe the effects of cardiopulmonary co-management on quality of life, symptoms and activity tolerance in subjects with COPD.
Change from baseline in CAT score in subjects with COPD. | Baseline,week4,week8,week12
  To describe the effects of cardiopulmonary co-management on quality of life, symptoms and activity tolerance in subjects with COPD.
Change from baseline in SGRQ score in subjects with COPD. | Baseline,week4,week8,week12
  To describe the effects of cardiopulmonary co-management on quality of life, symptoms and activity tolerance in subjects with COPD.
Change from baseline in 6MWD score in subjects with COPD. | Baseline,week4,week8,week12
  To describe the effects of cardiopulmonary co-management on quality of life, symptoms and activity tolerance in subjects with COPD.
Change from baseline in pre-dose FEV1 and FVC value | Baseline,week12
  To describe the effects of cardiopulmonary co-management on lung function in subjects with COPD.
Change from baseline in FEV1 and FVC value within 4 hours post-dosing. | Baseline,week12
  To describe the effects of cardiopulmonary co-management on lung function in subjects with COPD.
The rate of AF recurrence in subjects with AF and COPD. | Baseline-week12
  To describe the rate of AF recurrence during the period of cardiopulmonary co-management.
Change from baseline in BNP/NT-proBNP value in the subjects with CHF and COPD. | Baseline,week12
  To describe the change of biomarkers in the subjects with CVD and COPD during the period of cardiopulmonary co-management.
Change from baseline in blood lipids value(TC, LDL, HDL and TG) in the subjects with CHD and COPD. | Baseline,week12
  To describe the change of biomarkers in the subjects with CVD and COPD during the period of cardiopulmonary co-management.
Propotion of newly diagnosed COPD patients in subjects with COPD at baseline. | Baseline
  To describe the undiagnosed rate of COPD in subjects with CVD.
Propotion of newly diagnosed COPD patients in CHD, AF and CHF subjects with COPD at baseline. | Baseline
  To describe the undiagnosed rate of COPD in subjects with CVD.
Propotion of subjects at high risk of COPD in subjects with CVD, CHD, AF and CHF at baseline. | Baseline
  To describe the proportion of subjects at high risk of COPD among CVD patients.
Propotion of subjects at high risk of COPD diagnosed with COPD in subjects with CVD, CHD, AF and CHF at baseline. | Baseline
  To describe the proportion of subjects at high risk of COPD among CVD patients.
Distribution of stable COPD medications by drug class (ICS, ICS/LABA, methylxanthines,etc) and others [antibiotics, systemic corticosteroids, traditional Chinese medicine, etc]) in mono or combination at baseline and week 12. | Baseline,week12
  To describe the COPD-related treatment patterns before and after the implementation of cardiopulmonary co-management.

OTHER OUTCOMES:
The exacerbation rate in CVD, CHD, AF and CHF subjects with COPD over 12 weeks. | Baseline-week12
  To explore the exacerbation rate in subjects with CVD and COPD during the period of cardiopulmonary co-management.
Rate of MACE in CVD, CHD, AF and CHF subjects with COPD over 12 weeks. | Baseline-week12
  To explore the occurrence of MACE event in subjects with CVD and COPD during the period of cardiopulmonary co-management.
Rate of differente types of MACE in CVD, CHD, AF and CHF subjects with COPD over 12 weeks. | Baseline-week12
  To explore the occurrence of MACE event in subjects with CVD and COPD during the period of cardiopulmonary co-management.
Risk factors for COPD diagnosis in CHD, AF and CHF subjects (analysis scope includes demographics, physiological data, family history, smoking status, age, comorbidities, lung function parameters, biomarkers, etc.) | Baseline
  To explore the risk factors in CVD subjects with COPD.
Risk factors for MACE in subjects with CVD and COPD (analysis scope includes baseline characteristics, baseline PROs, drug treatment, non-drug treatment, lung function parameters, biomarkers, etc.) | Baseline
  To explore the risk factors of MACE in subjects with CVD and COPD.
Change(Mean, standard deviation, median, interquartile range, minimum, and maximum values) from baseline in pre-dose and post-dose IOS parameters(Z at 5 Hz [kPa/(L/s)]、R at 5 Hz [kPa/(L/s)]、R at 10 Hz [kPa/(L/s)] and so on) at week 12. | Baseline,week12
  To explore the changes in IOS parameters in subjects with COPD during the period of cardiopulmonary co-management.
Correlation(via Spearman's rank correlation coefficient(-1 to 1), -1=negative correlation,0=no correlation, +1=positive correlation) between change from baseline in pre-dose/post-dose IOS parameters and change from baseline in CAT score at week 12. | Baseline,week12
  To explore the correlation between changes in IOS parameters and symptoms in COPD subjects.
Correlation(via Spearman's rank correlation coefficient(-1 to 1), -1=negative correlation,0=no correlation, +1=positive correlation) between change from baseline in pre-dose/post-dose IOS parameters and change from baseline in mMRC score at week 12. | Baseline,week12
  To explore the correlation between changes in IOS parameters and symptoms in COPD subjects.
Correlation(via Spearman's rank correlation coefficient(-1 to 1), -1=negative correlation,0=no correlation, +1=positive correlation) between change from baseline in pre/post-dose spirometry parameters and change from baseline in CAT score at week 12. | Baseline,week12
  To explore the correlation between changes in spirometry parametersH and symptoms in COPD subjects.
Correlation(via Spearman's rank correlation coefficient(-1 to 1), -1=negative correlation,0=no correlation, +1=positive correlation) between change from baseline in pre/post-dose spirometry parameters and change from baseline in mMRC score at week 12. | Baseline,week12
  To explore the correlation between changes in spirometry parametersH and symptoms in COPD subjects.

CONTACTS AND LOCATIONS:
Locations (26):
- China (26):
  - Research Site, Beijing
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Dongguan
  - Research Site, Foshan
  - Research Site, Guangzhou
  - Research Site, Haikou
  - Research Site, Hubei
  - Research Site, Jiujiang
  - Research Site, Kaiyuan
  - Research Site, Kunming
  - Research Site, Leping
  - Research Site, Linhai
  - Research Site, Mianyang
  - Research Site, Nanchang
  - Research Site, Shanghai
  - Research Site, Shantou
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Shijiazhuang
  - Research Site, Suining
  - Research Site, Xi'an
  - Research Site, Xuzhou
  - Research Site, Yangzhou
  - Research Site, Zhengzhou
  - Research Site, Zunyi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. 'Yes' , indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/